CLINICAL TRIAL: NCT02808156
Title: Effectiveness of Unilateral Versus Bilateral Intensive Training in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201512070RINA
Record Dates: First submitted 2016-05-24; First posted 2016-06-21 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy,; Upper limb neurorehabilitation; Upper Extremity; Neurological Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- unilateral upper limbs intensive training (Experimental): The unimanual intensive training group focuses on the training of the more affected arm and restraint the less affected arm.
  Interventions: Other: unilateral upper limbs intensive training
- bilateral upper limbs intensive training (Experimental): The bimanual intensive training focuses activities that required the use of both hands.
  Interventions: Other: bilateral upper limbs intensive training

INTERVENTIONS:
Other: unilateral upper limbs intensive training — The unimanual intensive training group focuses on the training of the more affected arm and restraint the less affected arm.
  Arms: unilateral upper limbs intensive training
Other: bilateral upper limbs intensive training — The bimanual intensive training focuses activities that required the use of both hands.
  Arms: bilateral upper limbs intensive training

SUMMARY:
This 3-year research project aims to investigate and compare the immediate and long-term treatment effectiveness as well as motor improving curve and potential predictors of the unimanual intensive training and bimanual intensive training protocols with an equivalent intervention period in children with hemiplegic CP and children with CP with apparently one side affected. In addition, based on the ICF-CY model, comprehensive outcome measures including motor functions as well as psychological functions will be included.

ELIGIBILITY:
The inclusion criteria of this study are:

1. aged between 3 and 16 years
2. diagnosed with congenital hemiplegic or children with CP with one more affected side; (3) apparently disuse phenomenon of the more affected hand at spontaneous contexts

Participants will be exclude for:

1. excessive muscle tone (Modified Ashworth Scale ≤ 2 at any joints of the upper limb) before beginning treatment (Bohannon & Smith, 1987)
2. severe cognitive, visual, or auditory disorders according to medical documents, parental reports, and the examiner's clinical observation
3. injections of botulinum toxin type A or operations on the UE within 6 months

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes from Melbourne Assessment 2 (MA-2) | baseline, week 4, week 8, week 24
Changes from Pediatric Motor Activity Log-Revised (PMAL-R) | baseline, week 4, week 8, week 24
Changes from ABILHAND-Kids | baseline, week 4, week 8, week 24
Changes from Test of Playfulness (ToP) | week 1, week 4, week 5, week 8
Changes from Box and Block Test (BBT) | weekly test (from baseline to week 8)
Changes from Engagement Questionnaire (EQ) | weekly test (from week 1 to week 8)
Changes from Satisfactory Questionnaire (SQ) | baseline, week 4, week 8, week 24
Changes from Building Tower Test (BTT) | weekly test (from baseline to week 8)
Changes from String Beads Test (SBT) | weekly test (from baseline to week 8)
Changes from Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | baseline, week 4, week 8, week 24
Performance changes assessed by Kinematics Analysis | baseline, week 8, week 24
  Kinematic Analysis including parameters of endpoint control, inter-joints coordination, and trunk involvement, we will analyse children's performance changes from performing reaching tasks
Changes from muscle strength | baseline, week 8, week 24
  Measured by Electromyography (EMG)

SECONDARY OUTCOMES:
Changes from Pediatric Evaluation of Disability Inventory (PEDI) | baseline, week 4, week 8, week 24
Changes from Cerebral Palsy Quality of Life Questionnaire for Children (CPQOL) | baseline, week 4, week 8, week 24
Changes from Parenting Stress Index-Short Form (PSI-short) | baseline, week 4, week 8, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Ni Wang, Principal Investigator — Department of Occupational Therapy, School of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan